CLINICAL TRIAL: NCT01247831
Title: The Effect of Selective Laser Trabeculoplasty (SLT) on Ocular Rigidity
Acronym: SLT/ORA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Dr. Karin Pillunat, Principla Investigator, Technische Universität Dresden
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SLT/ORA/1
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Glaucoma
Keywords: glaucoma, selective laser trabeculoplasty, ocular rigidity
MeSH Terms: conditions — Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- glaucoma patients (Other): All of the patients treated with SLT need further IOP reduction for control of their glaucoma.
  Interventions: Procedure: Selective Laser Trabeculoplasty

INTERVENTIONS:
Procedure: Selective Laser Trabeculoplasty — 100 spots with an energy of 0,8 mJ are applied over 360° of the trabecular meshwork of glaucoma patients with a Q-switched 532 nm frequency doubled neodymium YAG Laser.
  Other Names: SLT; ORA

SUMMARY:
The purpose of this study is to examine the influence of selective laser trabeculoplasty (SLT) on ocular rigidity in glaucoma patients.

DETAILED DESCRIPTION:
Ocular Rigidity (corneal hysteresis and corneal resistance factor) is measured with the Ocular Response Analyzer (Reichert) before and 4 weeks after SLT (Q-switched 532 nm frequency doubled neodymium yttrium aluminium garnet laser with a spot size of 400 µm and a 3-ns pulse duration). The trabecular meshwork is treated with 100 spots over 360° and an energy of 0,8 mJ.

The purpose is to examine if selective laser trabeculoplasty changes ocular rigidity.

ELIGIBILITY:
Inclusion Criteria:

glaucoma patients (primary open angle glaucoma, ocular hypertension) over the age of 18 who need further IOP reduction to control their glaucoma

Exclusion Criteria:

other forms of glaucoma (angle closure, secondary glaucoma, congenital, juvenile), acute psychosis, epilepsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2010-11; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
change in ocular rigidity | 4 weeks
  Is there a change in ocular rigidity (corneal hysteresis, corneal resistance factor) as measured with the Ocular Response Analyzer (Reichert) after selective laser trabeculoplasty?

SECONDARY OUTCOMES:
IOP reduction | 4 weeks
  Is there an effective IOP drop after SLT?

CONTACTS AND LOCATIONS:
Overall Officials: Karin R Hornykewycz, MD, Principal Investigator — University Eye Clinic Dresden
Locations (1):
- University Eye Clinic Dresden, Dresden, Saxony, Germany